CLINICAL TRIAL: NCT02359643
Title: Multi-center Prospective Randomized Control Trail of High Dose Aspirin in Acute Stage of Kawasaki Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kawasaki Disease
Record Dates: First submitted 2015-01-05; First posted 2015-02-10 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2013-05

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with high dose aspirin (Placebo Comparator): KD patients treated with high dose IVIG (2gm/kg) and high dose aspirin (>50mg/kg/day) since diagnosed, then taper to low dose aspirin (3-5mg/kg/day) when fever subside.
  Interventions: Drug: Aspirin
- Without high dose aspirin (Experimental): KD patients treated with high dose IVIG (2gm/kg) without high dose aspirin (>50mg/kg/day) since diagnosed, then low dose aspirin (3-5mg/kg/day) when fever subside.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — This study was conduct to investigate the role of high dose aspirin in acute stage of KD via a multi-center randomized control trail, and we plan to achieve the followings in the coming 4 years:
  1. Enroll 300 KD patients from multiple medical centers of Taiwan and China in 4 years. Randomize group patients as group 1: with high dose aspirin (more than 30/mg/kd/day) until fever subsided and shift to low dose aspirin (3-5mg/kg/day, N=150); and group 2: without high dose aspirin during acute febrile stage, only use low dose aspirin (N=150).
  2. Compare data including fever days, admission duration, laboratory data (CBC/DC, GOT/GPT, BUN/Cr, Alb, ESR, CRP, 2D echo), IVIG treatment response and CAL formation rate (followed at least 1 year).
  Other Names: acetylsalicylic acid

SUMMARY:
Kawasaki disease (KD) is an acute multi-system vasculitis syndrome of unknown etiology occurring mostly in infants and children younger than 5 years of age. In developed countries, it is the leading cause of acquired heart disease in children. However, KD remains a mysterious disease.

Single high dose intravenous immunoglobulin (IVIG, 2gm/kg) and aspirin are standard treatment for KD. Aspirin have been prescribed in treatment of KD for decade even earlier than usage of IVIG. High dose aspirin mainly act as anti-inflammation, while low dose aspirin as anti-platelet. IVIG may play most of the role of anti-inflammation in acute stage of KD. Hsieh et al. reported that KD without high dose aspirin had the same treatment response after IVIG. Therefore it is still unclear about the necessarily of high dose aspirin in acute stage of KD.

This study was conduct to investigate the role of high dose aspirin in acute stage of KD via a multi-center randomized control trail, and we plan to achieve the followings till year 2017:

1. Enroll 300 KD patients from multiple medical centers . Randomize group patients as group 1: with high dose aspirin (more than 30/mg/kd/day) until fever subsided and shift to low dose aspirin (3-5mg/kg/day, N=150); and group 2: without high dose aspirin during acute febrile stage, only use low dose aspirin (N=150).
2. Compare data including fever days, admission duration, laboratory data (CBC/DC, GOT/GPT, BUN/Cr, Alb, ESR, CRP, 2D echo), IVIG treatment response and CAL formation rate (followed at least 1 year).

DETAILED DESCRIPTION:
All subjects are children who fulfilled the criteria for KD and who are treated with IVIG at each hospital after informed contents are obtained. The patients are initially treated with a single dose of IVIG (2 g/kg) during a 12-hour period.

Principal clinical features of KD that occur in the acute stage within 5 days of the onset of fever will be recorded. After the informed content from the parents, PB samples will be obtained before IVIG treatment (pre-IVIG, KD1), within 3 days after complete initial IVIG treatment (post-IVIG, KD2) as the acute stage samples and then 1 month, 6 month and 12 month followed-up as subacute/convalescent stage samples. CAL was defined as the internal diameter being at least 3 mm of the coronary artery (4 mm if the subject was over the age of 5 years) or the internal diameter of a segment at least 1.5 times as large as that of an adjacent segment by echocardiogram.

High dose aspirin will be given (> 30 mg/kg/day) until the fever subsided at group 1 randomly. After fever subside (<38C, for 48 hours) low-dose aspirin (3-5 mg/kg/day) will be prescribed for all patients until all signs of inflammation resolved in both group 1 and 2.

ELIGIBILITY:
Inclusion Criteria: (both 1 and 2)

1. All subjects are children who fulfilled the criteria for Kawasaki Disease (American Heart Association criteria).

1. Fever > 5 days, and 4 of the 5 following symptoms
2. Diffuse mucosal inflammation (strawberry tongue, dry and fissured lips)
3. Bilateral non-purulent conjunctivitis,
4. Dysmorphous skin rashes,
5. Indurative angioedema over the hands and feet
6. Cervical lymphadenopathy. (One or more nodule at lease 1.5 cm in diameter) 2. KD patients are treated with IVIG at each hospital after informed contents are obtained.

Exclusion Criteria:

1. Patients whose symptoms did not full fit the Kawasaki Disease criteria.
2. Had an acute fever for < 5 days and >10 days
3. Incomplete collection of each followed-up data (CBC/DC, GOT/GPT, BUN/Cr, Albumin, ESR, C-Reactive Protein, 2D echocardiography)
4. IVIG treatment at other hospital before refers to study centers.
5. Treatment with corticosteroids, other than inhaled forms, in the previous 2 weeks before enrollment;
6. The presence of a disease known to mimic Kawasaki disease.
7. Previous diagnosis of Kawasaki disease
8. Inability to take aspirin

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
To assess total hospital day | 5-10 days

SECONDARY OUTCOMES:
To assess total fever duration | 5-10 days
To assess how many times of intramenous immunoglobulin (IVIG) treatment | 21 days
  IVIG resistance: more than 2 times of IVIG (2gm/kg); or IVIG responsive: only treatment with one time of IVIG (2gm/kg)
To examine whether coronary artery lesion formation (CAL) | 6-8 weeks
  CAL was defined as the internal diameter being at least 3 mm of the coronary artery (4 mm if the subject was over the age of 5 yr) or the internal diameter of a segment at least 1.5 times as large as that of an adjacent segment by echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Chang Kuo, MD, PhD, Study Chair — Chang Gung Memorial Hospital

REFERENCES:
- [Background] Hsieh KS, Weng KP, Lin CC, Huang TC, Lee CL, Huang SM. Treatment of acute Kawasaki disease: aspirin's role in the febrile stage revisited. Pediatrics. 2004 Dec;114(6):e689-93. doi: 10.1542/peds.2004-1037. Epub 2004 Nov 15. PMID 15545617
- [Background] Chen CH, Lin LY, Yang KD, Hsieh KS, Kuo HC. Kawasaki disease with G6PD deficiency--report of one case and literature review. J Microbiol Immunol Infect. 2014 Jun;47(3):261-3. doi: 10.1016/j.jmii.2012.05.002. Epub 2012 Jun 23. PMID 22727889